CLINICAL TRIAL: NCT00828243
Title: Genetic Regulation of Surfactant Deficiency in Human Newborn Infants
Brief Title: Genetic Regulation of Surfactant Deficiency
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 07-0156; R01HL082747 (NIH)
Record Dates: First submitted 2009-01-22; First posted 2009-01-23 (Estimated); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Respiratory Distress Syndrome, Newborn
Keywords: Pulmonary surfactants; Pulmonary surfactant associated protein B; Pulmonary surfactant associated protein C; ATP-binding cassette protein sub member family A3
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn | interventions — Nutrients; Acetates; Leucine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA samples and tracheal aspirate samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Genetic association: Infants with and without neonatal respiratory distress syndrome undergo surfactant gene sequencing to identify genomic variants associated with neonatal respiratory distress syndrome
- Nutrient: To newborn infants with respiratory distress syndrome, we administer stable isotopically labeled nutrients (precursors of surfactant phospholipids or proteins) to permit mass spectrometry-based comparison of surfactant phospholipid and protein turnover.
  Interventions: Drug: Nutrient

INTERVENTIONS:
Drug: Nutrient — We administer stable isotopically labeled precursors of surfactant phospholipids ([1-13C1] acetate) and of surfactant protein-B ([5,5,5-2H3] leucine) to infants with neonatal respiratory distress syndrome. Using mass spectrometry, we measure incorporation of stable isotopically labeled precursors in tracheal aspirates and compare surfactant phospholipid and surfactant protein-B turnover.
  Other Names: [1-13C1] acetate, [5,5,5-2H3] leucine
  Groups: Nutrient

SUMMARY:
Inherited deficiencies in any one of 3 genes (surfactant protein B, surfactant protein C, and ATP-binding cassette transporter A3) can cause neonatal respiratory distress syndrome by disrupting metabolism of the pulmonary surfactant. The investigators will use state of the art methods to link specific changes in the genetic code of each of these genes with disruption of discrete steps in the metabolism of the pulmonary surfactant in human newborn infants. These studies will lead to improved diagnostic capabilities and suggest novel strategies to correct surfactant deficiency in newborn infants.

DETAILED DESCRIPTION:
Genetic regulation of neonatal pulmonary surfactant deficiency has been suggested by studies of gender, genetic linkage, recurrent familial cases, targeted gene ablation in murine lineages, and by racial disparity in risk of neonatal respiratory distress syndrome. Successful fetal-neonatal pulmonary transition requires production of the pulmonary surfactant, a phospholipid-protein film that lines alveoli and maintains alveolar patency at end expiration. Our goal is to understand the genetic mechanisms that disrupt pulmonary surfactant metabolism and cause neonatal respiratory distress syndrome. Studies in human newborn infants have demonstrated that 3 genes are critical for surfactant metabolism: surfactant protein B (SFTPB), surfactant protein C (SFTPC), and an ATP-binding cassette transporter, ABCA3 (ABCA3). To understand genetic regulatory mechanisms, we will investigate the contribution of variation in each of these genes to risk of neonatal respiratory distress syndrome by testing the hypothesis that genetic variants in the SFTPB, SFTPC, and ABCA3 disrupt pulmonary surfactant metabolism. Using high throughput automated sequencing to genotype, multidimensional protein identification technology to assess quantitative and qualitative differences in surfactant protein B and C expression, in vivo metabolic labeling with stable isotopically labeled precursors to estimate surfactant protein B and C and phospholipid metabolic rates, and cohort sizes that provide statistical power (0.8), we will use race-specific, severity-stratified case-control (N=480) and case comparison (N=250) designs to understand genetically regulated, metabolic mechanisms that cause surfactant deficiency by disrupting expression or altering processing of surfactant proteins B or C or by disrupting surfactant phospholipid composition in human newborn infants. Improved understanding of genetic regulation of surfactant deficiency will suggest novel diagnostic strategies to identify and categorize high risk infants and therapeutic strategies that target discrete steps in pulmonary surfactant metabolism to improve outcomes of infants with neonatal respiratory distress syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Newborn infants with respiratory distress syndrome who require mechanical ventilation via endotracheal tube or tracheostomy in the first 6 months of life

Exclusion Criteria:

* Infants with conditions likely to cause imminent death

Ages: 1 Day to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population includes infants with and without neonatal respiratory distress syndrome (N=513) and infants with varying severity of neonatal respiratory distress syndrome (N=12).
Sampling Method: Non-Probability Sample
Enrollment: 525 (Actual)
Dates: Start 2007-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Association of specific variants or interactions among variants in SFTPB, SFTPC, and ABCA3 with neonatal respiratory distress syndrome | 1 week
  Statistical association of increased risk of neonatal respiratory distress in term or near term infants with specific genomic variants in SFTPB, SFTPC, and ABCA3

SECONDARY OUTCOMES:
Association of specific variants or interactions among variants in SFTPB, SFTPC, and ABCA3 with fractional synthetic rate and/or fractional catabolic rate of surfactant phospholipids, surfactant protein-B, and surfactant protein-C | 1 week
  Statistical association of quantitative surfactant phospholipid metabolic characteristics with specific genomic variants in SFTPB, SFTPC, and ABCA3

CONTACTS AND LOCATIONS:
Overall Officials: F. S. Cole, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- St. Louis Children's Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
Enter discovered genomic variants in dbGaP

REFERENCES:
- [Background] Tomazela DM, Patterson BW, Hanson E, Spence KL, Kanion TB, Salinger DH, Vicini P, Barret H, Heins HB, Cole FS, Hamvas A, MacCoss MJ. Measurement of human surfactant protein-B turnover in vivo from tracheal aspirates using targeted proteomics. Anal Chem. 2010 Mar 15;82(6):2561-7. doi: 10.1021/ac1001433. PMID 20178338
- [Background] Hamvas A, Heins HB, Guttentag SH, Wegner DJ, Trusgnich MA, Bennet KW, Yang P, Carlson CS, An P, Cole FS. Developmental and genetic regulation of human surfactant protein B in vivo. Neonatology. 2009;95(2):117-24. doi: 10.1159/000153095. Epub 2008 Sep 6. PMID 18776725
- [Result] Hamvas A, Nogee LM, Wegner DJ, Depass K, Christodoulou J, Bennetts B, McQuade LR, Gray PH, Deterding RR, Carroll TR, Kammesheidt A, Kasch LM, Kulkarni S, Cole FS. Inherited surfactant deficiency caused by uniparental disomy of rare mutations in the surfactant protein-B and ATP binding cassette, subfamily a, member 3 genes. J Pediatr. 2009 Dec;155(6):854-859.e1. doi: 10.1016/j.jpeds.2009.06.006. Epub 2009 Aug 3. PMID 19647838
- [Result] McBee AD, Wegner DJ, Carlson CS, Wambach JA, Yang P, Heins HB, Saugstad OD, Trusgnich MA, Watkins-Torry J, Nogee LM, Henderson H, Cole FS, Hamvas A. Recombination as a mechanism for sporadic mutation in the surfactant protein-C gene. Pediatr Pulmonol. 2008 May;43(5):443-50. doi: 10.1002/ppul.20782. PMID 18383112
- [Result] Garmany TH, Wambach JA, Heins HB, Watkins-Torry JM, Wegner DJ, Bennet K, An P, Land G, Saugstad OD, Henderson H, Nogee LM, Cole FS, Hamvas A. Population and disease-based prevalence of the common mutations associated with surfactant deficiency. Pediatr Res. 2008 Jun;63(6):645-9. doi: 10.1203/PDR.0b013e31816fdbeb. PMID 18317237
- [Result] Wambach JA, Yang P, Wegner DJ, An P, Hackett BP, Cole FS, Hamvas A. Surfactant protein-C promoter variants associated with neonatal respiratory distress syndrome reduce transcription. Pediatr Res. 2010 Sep;68(3):216-20. doi: 10.1203/PDR.0b013e3181eb5d68. PMID 20539253
- [Result] Anadkat JS, Kuzniewicz MW, Chaudhari BP, Cole FS, Hamvas A. Increased risk for respiratory distress among white, male, late preterm and term infants. J Perinatol. 2012 Oct;32(10):780-5. doi: 10.1038/jp.2011.191. Epub 2012 Jan 5. PMID 22222548
- [Result] Agrawal A, Hamvas A, Cole FS, Wambach JA, Wegner D, Coghill C, Harrison K, Nogee LM. An intronic ABCA3 mutation that is responsible for respiratory disease. Pediatr Res. 2012 Jun;71(6):633-7. doi: 10.1038/pr.2012.21. Epub 2012 Feb 15. PMID 22337229
- [Result] Bereman MS, Tomazela DM, Heins HS, Simonato M, Cogo PE, Hamvas A, Patterson BW, Cole FS, MacCoss MJ. A method to determine the kinetics of multiple proteins in human infants with respiratory distress syndrome. Anal Bioanal Chem. 2012 Jun;403(8):2397-402. doi: 10.1007/s00216-012-5953-3. Epub 2012 Apr 14. PMID 22526637
- [Result] Wambach JA, Wegner DJ, Depass K, Heins H, Druley TE, Mitra RD, An P, Zhang Q, Nogee LM, Cole FS, Hamvas A. Single ABCA3 mutations increase risk for neonatal respiratory distress syndrome. Pediatrics. 2012 Dec;130(6):e1575-82. doi: 10.1542/peds.2012-0918. Epub 2012 Nov 19. PMID 23166334
- [Result] Wambach JA, Wegner DJ, Heins HB, Druley TE, Mitra RD, Hamvas A, Cole FS. Synonymous ABCA3 variants do not increase risk for neonatal respiratory distress syndrome. J Pediatr. 2014 Jun;164(6):1316-21.e3. doi: 10.1016/j.jpeds.2014.02.021. Epub 2014 Mar 20. PMID 24657120
- [Result] Wambach JA, Casey AM, Fishman MP, Wegner DJ, Wert SE, Cole FS, Hamvas A, Nogee LM. Genotype-phenotype correlations for infants and children with ABCA3 deficiency. Am J Respir Crit Care Med. 2014 Jun 15;189(12):1538-43. doi: 10.1164/rccm.201402-0342OC. PMID 24871971
- [Result] Jackson T, Wegner DJ, White FV, Hamvas A, Cole FS, Wambach JA. Respiratory failure in a term infant with cis and trans mutations in ABCA3. J Perinatol. 2015 Mar;35(3):231-2. doi: 10.1038/jp.2014.236. PMID 25712598